CLINICAL TRIAL: NCT02871076
Title: Acupuncture for Post-Traumatic Stress in Combat Veterans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southern California Institute for Research and Education (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Hollifield, MD, Director, Program for Traumatic Stress, Southern California Institute for Research and Education
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR151974
Record Dates: First submitted 2016-08-08; First posted 2016-08-18 (Estimated); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: PTSD; Acupuncture; Combat
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum Acupuncture (Experimental): Patients will receive verum acupuncture twice weekly for twelve weeks.
  Interventions: Device: Acupuncture
- Sham Placebo Acupuncture (Placebo Comparator): Patients will receive sham placebo acupuncture twice weekly for twelve weeks.
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture — Patients will be randomized to either treatment arm, verum acupuncture or sham placebo acupuncture.

SUMMARY:
The objective of this study is to determine if acupuncture is an effective treatment option for treating combat Veterans with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Veteran Age 18 to 55
* DSM-5 criteria for chronic PTSD on Clinical Administered PTSD Scale (CAPS-5)
* CAPS-5 score of ≥ 26 and meeting criteria for each of 4 symptoms

Exclusion Criteria:

* Current and past six-months psychosis
* Substance dependence within 6 months (evidence of tolerance and/or withdrawal)
* Thyroid disease
* Decisional incapacity (e.g., dementia)
* Centrally acting medications that have a potential effect on biological expression (e.g., beta-blockers, opiates, and ≥10mg equivalent of diazepam/day)
* Pain levels requiring opiate medications
* Known exposure to chemicals or physical trauma that cause neuropsychiatric sequelae
* Severe depression (Beck Depression Inventory-II score ≥30)
* A diagnosed and untreated sleep breathing disorder (SBD)
* High risk of a SBD as indicated by snoring ≥50 of nights plus one of any

  1. Any witnessed apnea
  2. Feeling non-refreshed in the morning ≥50 of mornings
  3. Daytime sleepiness indicated by falling asleep with routine tasks such as watching TV or reading
* Non-response to ≥2 evidence-based PTSD treatments (adequate medication of 12 weeks or completion to PE, CPT or an intensive program)
* Treatment non-adherence indicated by stopping treatment or >3 missed appointments in the course of PTSD EBT
* High dissociation as indicated by a score of ≥25 on the Dissociative Experiences Scale - II
* Past chronic PTSD prior to military service
* Current active psychotherapy for PTSD
* Having acupuncture in the past year
* Pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-05-19 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Clinician Administered PTSD Scale (CAPS-5) PTSD Diagnosis | 4 months: Baseline CAPS to post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hollifield, MD, Principal Investigator — Tibor Rubin VA Medical Center
Locations (1):
- Veterans Affairs Long Beach Healthcare System, Long Beach, California, United States